CLINICAL TRIAL: NCT00976222
Title: Intravitreal Ranibizumab in Patients With Retinal Pigment Epithelial Detachments Secondary to Age-related Macular Degeneration
Brief Title: Intravitreal Ranibizumab in Retinal Pigment Epithelial Detachments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Nicole Eter, Director of Ophthalmology Department, University Hospital Muenster
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD-PED 08; Eudra-CT: 2008-004675-22
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Pigment Epithelial Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Intravitreal Injections; Ranibizumab

ARMS (1):
- 1 Arm Ranibizumab (Other)
  Interventions: Drug: intravitreal injection with ranibizumab

INTERVENTIONS:
Drug: intravitreal injection with ranibizumab — 0.5 mg in 0.05 ml, monthly, 12 months
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to demonstrate the efficacy of ranibizumab in patients with retinal pigment epithelial detachment secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Pigment epithelial detachments (PED) secondary to age-related macular degeneration (AMD) have been excluded from practically all study populations of ranibizumab studies so far. PED represents a special entity in AMD. As yet, no standard treatment has been established for this disease.The stimuli that induce PED are not very well known, but there is evidence suggesting that angiogenic factors such as vascular endothelial growth factor (VEGF) also play a role in the pathogenesis. Ranibizumab is an anti-VEGF antibody fragment that blocks VEGF activity in patients with neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* patients with age-related macular degeneration and serous pigment epithelial detachment as determined by fluorescein and indocyanine green angiography and optical coherence tomography (OCT)
* patients who have a best-corrected visual acuity (BCVA) score between 73 and 24 ETDRS letters
* patients with pigment epithelial detachment (PED) ≥ 200 µm as determined by OCT
* male or female patients 50 years of age or greater
* patients willing and able to comply with all study procedures

Exclusion Criteria:

* patients with best-corrected visual acuity (BCVA) < 24 or >73 letters in the study eye
* patients previously treated by intravitreal injections of steroids or anti-VEGF agents, or patients previously treated by Verteporfin photodynamic therapy or focal laser photocoagulation
* history of uncontrolled glaucoma in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of ranibizumab in patients with retinal pigment epithelial detachment secondary to age-related macular degeneration | 12 months

SECONDARY OUTCOMES:
Safety | 12 months
Mean change in best corrected visual acuity | 12 months
Change in retinal thickness and height of pigment epithelial detachment | 12 months
Central visual field and stability of fixation | 12 months
Fluorescein leakage and changes in autofluorescence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Eter, MD, Principal Investigator — Dept. of Ophthalmology, University of Muenster Medical Center
Locations (2):
- Germany (2):
  - University Hospital Muenchen, München
  - University Hospital Muenster, Münster

REFERENCES:
- [Derived] Clemens CR, Wolf A, Alten F, Milojcic C, Heiduschka P, Eter N. Response of vascular pigment epithelium detachment due to age-related macular degeneration to monthly treatment with ranibizumab: the prospective, multicentre RECOVER study. Acta Ophthalmol. 2017 Nov;95(7):683-689. doi: 10.1111/aos.13359. Epub 2017 Jan 13. PMID 28084038